CLINICAL TRIAL: NCT04045652
Title: Modifiable Factors Predicting Persistence of Oncogenic HPV and Cervical Dysplasia in HIV Infected Kenyan Women
Brief Title: Factors Predicting Persistence of Oncogenic HPV and Cervical Dysplasia in HIV Infected Kenyan Women
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Patrick Joseph Loehrer Sr., Distinguished Professor of Medicine, Indiana University
Other Study IDs: IUCRO-0492
Record Dates: First submitted 2019-07-08; First posted 2019-08-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: HIV/AIDS; Cervical Dysplasia; HIV Infections
Keywords: HPV; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Uterine Cervical Dysplasia; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical and vaginal swabs Oral rinse or anal swab samples Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kenyan women: Kenyan women, some HIV-infected and some HIV-uninfected, VIA negative at enrollment.

SUMMARY:
This study will utilize a longitudinal study design to better understand the natural history of oncogenic Human Papillomavirus (HPV) infections in Human Immunodeficiency Virus (HIV)-infected and HIV-uninfected Kenyan women, including the potentially modifiable (and non-modifiable) factors that are associated with progression of oncogenic HPV infection to clinical disease, including cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Kenyan women who present for a cervical cancer screening at AMPATH-cervical cancer screening clinics at MTRH or Webuye and living in or within 30 km of the respective clinic at the time of informed consent
2. Between the ages of 18 -45 years old at the time of informed consent
3. Ability to provide written informed consent and HIPAA authorization
4. Must have a normal VIA
5. Must be willing and able to come to the clinic for visits and return for a 4 year follow-up visit

Exclusion Criteria:

1. History of an abnormal VIA or Pap smear
2. Diagnosis of CIN or cervical cancer
3. Signs or symptoms of a sexually transmitted infection (STI)
4. Women who are currently pregnant
5. Inability to understand and provide written informed consent due to a mental or physical disability, or a medical illness that has rendered the patient unable to understand consent or attend quarterly visits

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected and uninfected Kenyan women (age 18-45) living in or close to Eldoret who present to the AMPATH Cervical Cancer Screening Program (CCSP), at the Moi Referral and Teaching Hospital in Eldoret, Kenya for a cervical cancer screening will be asked if they would like information about this study.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Frequency of oncogenic Human Papillomavirus (HPV) in Human Immunodeficiency Virus(HIV)-infected women with a normal Visual Inspection with Acetic Acid (VIA) at baseline | Change in diagnosis from Baseline,months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  HPV testing will occur through cervical swabs for HPV and CT/GC testing, cervical VIA, as well as HPV swab (anal, cervical) and rinse samples (oral)
Frequency oncogenic HPV in non HIV-infected women with a normal VIA at baseline | change in diagnosis from Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up(1 year after the last visit)
  HPV testing will occur through cervical swabs for HPV and CT/GC testing, cervical VIA, as well as HPV swab (anal, cervical) and rinse samples (oral)
Incidence of abnormal VIA | Baseline

SECONDARY OUTCOMES:
Incidence of cervical dysplasia in Kenyan women with normal VIA at baseline, and who are HIV-infected during 4 years of observation | Incidence at Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  cervical and/or vaginal swabs for HPV and CT/GC testing
Incidence of cervical dysplasia in Kenyan women with normal VIA at baseline, and who are HIV-uninfected during 4 years of observation | Incidence at Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  cervical and/or vaginal swabs for HPV and CT/GC testing
Identify potentially modifiable sex behavioral risk factors associated with oncogenic HPV | Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  Through interviews/questionnaires
Identify potentially modifiable sex behavioral risk factors associated with cervical dysplasia | Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  Through interviews/questionnaires
Identify potentially modifiable health behavioral risk factors associated with oncogenic HPV | Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  Through interviews/questionnaires
Identify potentially modifiable health behavioral risk factors associated with cervical dysplasia | Baseline, months: 3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  Through interviews/questionnaires
Incidence of potentially modifiable biological risk factors associated with oncogenic HPV through HPV testing will occur through cervical and/or vaginal swabs | Baseline, months:3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  HPV testing will occur through cervical and/or vaginal swabs
Incidence of potentially modifiable biological behavioral risk factors associated with cervical dysplasia through cervical and/or vaginal swabs for HPV and CT/GC testing | Baseline, months:3,6,9,12,15,18,21,24,27,30,33,36,39,42,45,48 and follow-up (1 year after the last visit)
  cervical and/or vaginal swabs for HPV and CT/GC testing
Time to HPV | Baseline to HPV diagnosis (up to 2 years)
Time to Cervical Dysplasia | HPV diagnosis to Cervical Dysplasia (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (3):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States
- Moi University School of Medicine, Eldoret, Kenya
- Infectious Disease Institute, Makerere University, Kampala, Uganda